CLINICAL TRIAL: NCT04140500
Title: An Open Label, Multicenter, Dose Escalation, Phase 1 Study to Evaluate Safety/Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Anti Tumor Activity of RO7247669, a PD1-LAG3 Bispecific Antibody, in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: Dose Escalation Study of a PD1-LAG3 Bispecific Antibody in Patients With Advanced and/or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP41300; 2019-000779-18 (EudraCT Number)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors; Metastatic Melanoma; Non-small Cell Lung Cancer; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single-Agent Dose Escalation (Experimental): Participants will receive RO7247669 every 2 weeks (Q2W) or every 3 weeks (Q3W) up to the maximum tolerated dose (MTD) until disease progression, unacceptable drug toxicity, or withdrawal of consent, for up to 24 months.
  Interventions: Drug: RO7247669
- Part B: Tumor Specific Expansion Cohorts (Experimental): Participants with selected solid tumor indications will receive RO7247669 at a dose derived from Part A until disease progression, unacceptable drug toxicity, or withdrawal of consent, for up to 24 months.
  Interventions: Drug: RO7247669

INTERVENTIONS:
Drug: RO7247669 — Participants will receive intravenous (IV) RO7247669 at different doses either every 2 weeks (Q2W) or every 3 weeks (Q3W)

SUMMARY:
This is a first-in-human, open-label, multicenter, Phase I multiple-ascending dose (MAD) study of RO7247669, an anti PD-1 (programmed death-1) and LAG-3 (Lymphocyte-activation gene 3) bispecific antibody, for participants with advanced and/or metastatic solid tumors. This study aims to establish the maximum tolerated dose (MTD) and/or define the recommended phase 2 dose (RP2D) based on the safety, tolerability, pharmacokinetic (PK) and/or pharmacodynamic (PD) profile of RO7247669, and to evaluate preliminary anti-tumor activity in participants with solid tumors. An expansion part of the study is planned to enroll tumor-specific cohorts to evaluate anti-tumor activity of the MTD and/or RP2D of RO7247669 and to confirm safety and tolerability in participants with selected tumor types.

ELIGIBILITY:
Inclusion criteria

* Patient must have histologically or cytologically confirmed advanced and/or metastatic solid tumor malignancies for which standard curative or palliative measures do not exist, are no longer effective, or are not acceptable to the patient
* Eastern Cooperative Oncology Group Performance Status 0-1
* Fresh biopsies may be required
* Women of childbearing potential and male participants must agree to remain abstinent or use contraceptive methods as defined by the protocol

Additional Specific Inclusion Criteria for Participants with Melanoma

* Histologically confirmed, unresectable stage III or stage IV melanoma
* Not more than 2 prior lines of treatment for metastatic disease are allowed prior to enrolling in the study
* Prior treatment with an approved anti-PD-1 or anti-PD-L1 agent

Additional Specific Inclusion Criteria for Participants with Non-Small Cell Lung Cancer who Previously Received Treatment for Metastatic Disease

* Participants with histologically confirmed advanced non-small cell lung cancer
* Not more than 2 prior lines of treatment for metastatic disease are allowed prior to enrolling in the study
* Previously treated with approved PD-L1/PD-1 inhibitors
* Tumor PD-L1 expression as determined by immunohistochemistry assay of archival tumor tissue or tissue obtained at screening

Additional Specific Inclusion Criteria for Participants with Esophageal Squamous Cell Carcinoma

* Participants whose major lesion was histologically confirmed as squamous cell carcinoma or adenosquamous cell carcinoma of the esophagus
* Participants who have previously received not more than 1 prior line of treatment for metastatic disease prior to enrolling in the study

Additional Specific Inclusion Criteria for Participants with Non-Small Cell Lung Cancer who Previously did not Receive Treatment for Metastatic Disease

* Participants with histologically confirmed advanced non-small cell lung cancer
* Tumor PD-L1 expression as determined by immunohistochemistry assay of archival tumor tissue or tissue obtained at screening

Exclusion criteria

* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to any of the components of RO7247669
* Active or untreated central nervous system (CNS) metastases
* An active second malignancy
* Evidence of concomitant diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk from treatment complications
* Positive HIV, hepatitis B, or hepatitis C test result
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infection
* Vaccination with live vaccines within 28 days prior to Cycle 1 Day 1
* Treatment with oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* Active or history of autoimmune disease or immune deficiency
* Prior treatment with adoptive cell therapies, such as CAR-T therapies
* Concurrent therapy with any other investigational drug < 28 days or 5 half-lives of the drug, whichever is shorter, prior to the first RO7247669 administration
* Regular immunosuppressive therapy
* Radiotherapy within the last 4 weeks before start of study drug treatment, with the exception of limited palliative radiotherapy
* Prior treatment with a lymphocyte activation gene-3 (LAG-3) inhibitor

Additional Specific Exclusion Criteria for Participants with Non-Small Cell Lung Cancer who Previously Received Treatment for Metastatic Disease

* Participants with the following muations, rearrangements, translocations are not eligible: EGFR, ALK, ROS1, BRAFV600E, and NTRK

Additional Specific Exclusion Criteria for Participants with Esophageal Squamous Cell Carcinoma

* Prior therapy with any immunomodulatory agents

Additional Specific Exclusion Criteria for Participants with Non-Small Cell Lung Cancer who Previously did not Receive Treatment for Metastatic Disease

* Prior therapy for metastatic disease is not permitted
* Neo-adjuvant anti-PD-1 or anti-PD-L1 therapy is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Days 1-21 (Q2W dosing) or Days 1-28 (Q3W dosing) of Cycle 1
Part A: Percentage of Participants with Adverse Events | Baseline through the end of study (up to 24 months)
Part B: Objective Response Rate (ORR) | Up to 24 months
Part B: Disease Control Rate (DCR), Defined as ORR + Stable Disease Rate (SDR) | Up to 24 months
Part B: Duration of Response (DOR) | Up to 24 months
Part B: Progression-free Survival (PFS), Defined as the Time from the First Study Treatment to the First Occurrence of Progression per Investigator Assessment or Death from any Cause, Whichever Occurs First | Up to 24 months

SECONDARY OUTCOMES:
Parts A and B: Maximum Concentration (Cmax) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Time of Maximum Concentration (Tmax) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Clearance (CL) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Volume of Distribution at Steady State (Vss) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Area Under the Curve (AUC) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Half-Life (T1/2) of RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Parts A and B: Percentage of Participants with Anti-Drug Antibodies (ADA) to RO7247669 | Day 1 of each Cycle, starting with Cycle 1, through final study visit (up to 24 months)
Part B: Change from Baseline in T-Cell Activity | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Part A: Percentage of Receptors Occupied by RO7247669 | At pre-defined intervals from Day 1 of Cycle 1 through final study visit (up to 24 months)
Part A: ORR | At pre-defined intervals from initial dose up to 24 months
Part A: DCR | At pre-defined intervals from initial dose up to 24 months
Part A: PFS | At pre-defined intervals from initial dose up to 24 months
Part A: DOR | At pre-defined intervals from initial dose up to 24 months
Part B: Percentage of Participants with Adverse Events | Baseline through the end of study (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Denmark (2):
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- LLC Arensia Explorer Medicine, Tbilisi, Georgia
- Israel (3):
  - Hadassah University Hospital - Ein Kerem, Jerusaelm
  - Rabin MC, Petah Tikva
  - Chaim Sheba medical center, Oncology division, Ramat Gan
- Mexico (3):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Inst. Nacional de Cancerología, Mexico City, Mexico CITY (federal District)
  - Consultorio Médico Jordi Guzmán Casta, Querétaro City, Querétaro
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
- Turkey (Türkiye) (4):
  - Adana City Hospital, Medical Oncology, Adana
  - Ankara City Hospital, Ankara
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara
  - Ankara Abdurrahman Yurtaslan Oncology Training and Research Hospital Phase 1 Center, Yen?mahalle
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Christie Hospital NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing